CLINICAL TRIAL: NCT07333209
Title: Determine the Impact of Scheduled Positioning With a Peanutball on Labor Outcomes Among Primiparous Women Under Epidural Analgesia: A Non-Invasive Randomized Controlled Trial
Brief Title: Scheduled Positioning With a Peanutball(SPP) on Labor Outcomes Among Primiparous Women Under Epidural Analgesia
Acronym: Peanutball
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Ms. Parveen Nather, Principal Investigator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MRC-01-25-1104
Record Dates: First submitted 2025-12-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Labor (Obstetrics)--Complications
Keywords: Peanutball; Scheduled positioning; Primiparous women; Randomized controlled trial; Non-invasive intrapartum intervention; Maternal labor outcomes; Neonatal outcomes; Epidural Analgesia

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group randomized controlled trial design in which primigravida women receiving epidural analgesia are randomly assigned to either an intervention group-receiving scheduled maternal position changes using a peanut birthing ball-or a control group receiving standard intrapartum care without the peanut ball. Outcomes for both groups will be compared prospectively to determine the effect of the intervention on labor progression and maternal and neonatal outcomes.
Who Masked: Outcomes Assessor
Masking Description: This study is assessor-blinded. Due to the nature of the intervention (scheduled maternal positioning using a peanut ball), participants, care providers, and investigators are not masked, as the intervention is visible and requires active participation in care.
  The outcomes assessor is masked to group assignment and does not participate in the delivery of the intervention. Outcome data are collected using standardized tools and extracted from medical records without indication of whether the participant received the peanut ball intervention or standard care, in order to minimize assessment bias. No other parties masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Peanut Ball-Assisted Scheduled Maternal Positioning
  Interventions: Other: Scheduled Maternal Positioning with use of peanutball
- Control Arm (Active Comparator): Standard Intrapartum Care
  Interventions: Other: Scheduled Maternal Positioning with use of peanutball

INTERVENTIONS:
Other: Scheduled Maternal Positioning with use of peanutball — Participants will receive standard intrapartum care following epidural analgesia plus scheduled maternal position changes using a peanut birthing ball. The peanut ball will be placed between the participant's legs, and maternal positions will be changed at predefined intervals according to the study protocol. Positions include left lateral, right lateral, semi-sitting, and Taylor positions. All positioning will be supervised by trained nursing and midwifery staff and adjusted as needed based on maternal comfort and fetal heart rate monitoring.

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate whether scheduled maternal position changes using a peanut birthing ball improve labor outcomes in low-risk, primiparous women receiving epidural analgesia during labor. The main questions it aims to answer are:

Does scheduled maternal positioning with a peanut ball reduce the duration of the first and second stages of labor?

Does scheduled maternal positioning with a peanut ball influence mode of delivery and maternal and neonatal outcomes?

This non-invasive randomized controlled trial will be conducted at the Women's Wellness and Research Center in Qatar. Participants will be randomly assigned to either an intervention group receiving scheduled maternal position changes using a peanut birthing ball or a control group receiving standard intrapartum care without peanut ball use. Researchers will compare outcomes between the two groups to determine whether structured positioning with a peanut ball improves labor progression and delivery outcomes in women receiving epidural analgesia.

Participants in the intervention group will undergo scheduled position changes throughout labor using a peanut birthing ball, including left lateral, right lateral, semi-sitting, and Taylor positions, under the supervision of trained nursing and midwifery staff. Participants in the control group will receive routine intrapartum care following epidural analgesia without the use of a peanut ball or a structured positioning schedule.

Primary maternal outcomes include duration of the first and second stages of labor, mode of delivery, estimated blood loss, postpartum hemorrhage, use of oxytocin augmentation, degree of perineal trauma, and hospitalization cost. Neonatal outcomes include Apgar scores at 5 and 10 minutes, NICU admission, birth-related injuries, and umbilical cord blood pH. Findings from this study are expected to support evidence-based intrapartum care practices and inform clinical protocols for women receiving epidural analgesia.

DETAILED DESCRIPTION:
1. Background and Introduction

   Labor pain is recognized as one of the most intense forms of physiological pain experienced in human medicine. Although pain during childbirth is a natural and expected process, contemporary evidence-based practice supports the provision of pain relief upon maternal request, with maternal preference for analgesia considered a sufficient clinical indication. Epidural analgesia (EA) is widely regarded as the most effective pharmacological method for labor pain relief. By administering local anesthetic agents into the epidural space, EA produces a dense sensory block of the lower abdomen and lower extremities, significantly reducing or abolishing labor pain while generally preserving maternal consciousness and cooperation.

   Globally, the use of epidural analgesia during labor varies but is particularly common in high-resource healthcare settings. Utilization rates range from approximately 20% to 80% of laboring women, with national estimates indicating use in around 67% of parturients in the United States, 60% in the United Kingdom, and nearly 80% in France. Despite high maternal satisfaction and effective pain control, epidural analgesia has been associated in some studies with prolonged labor, particularly during the first and second stages, and with increased rates of instrumental vaginal delivery and cesarean section. These associations remain a subject of ongoing clinical and research debate.

   The World Health Organization (WHO) emphasizes maternal mobility and optimal positioning during labor as essential strategies to promote physiological birth, facilitate fetal descent, and reduce unnecessary obstetric interventions. However, in routine clinical practice, women receiving epidural analgesia frequently experience restricted mobility due to partial motor blockade, continuous fetal heart rate monitoring, and bed confinement. These factors limit the use of upright and gravity-assisted positions that may otherwise support labor progress and optimal fetal positioning.
2. Maternal Labor Positions and Peanut Ball Use

Multiple maternal positions are recommended during labor to optimize uteroplacental perfusion, encourage fetal rotation, and enhance maternal comfort. These include lateral positions, semi-sitting postures, and modified sitting positions such as the Taylor position.

The left lateral position reduces aortocaval compression, improves uteroplacental blood flow, enhances fetal oxygenation, and may facilitate rotation of the fetus from occiput posterior to occiput anterior. The right lateral position provides similar physiological benefits while preventing prolonged pressure on one side. Semi-sitting or semi-reclining positions utilize gravity to assist fetal engagement and may shorten the second stage of labor. The Taylor (modified sitting) position increases the subpubic angle and pelvic outlet diameter, promoting fetal descent and spontaneous vaginal birth.

Birthing balls have emerged as low-cost, non-pharmacological interventions to support physiological labor. Among these, the peanut birthing ball-a peanut-shaped inflatable device placed between the thighs or knees-has gained popularity, particularly among women receiving epidural analgesia who have limited mobility. The peanut ball facilitates hip abduction, widens pelvic dimensions, maintains optimal spinal alignment, and simulates upright or squatting positions while allowing the woman to remain in bed.

Several randomized controlled trials have examined the impact of peanut ball use during labor, reporting potential benefits such as reduced duration of labor, improved cervical dilation, higher rates of spontaneous vaginal birth, and reduced primary cesarean delivery. However, systematic reviews and meta-analyses have reported inconsistent findings, with some demonstrating benefit and others showing no statistically significant differences compared with standard care.

3. Evidence Gaps and Rationale

Recent systematic reviews and meta-analyses highlight significant heterogeneity in peanut ball intervention protocols, including variations in positioning type, frequency, duration, and timing. Many studies rely on unsystematic or clinician-driven repositioning rather than standardized schedules, limiting the ability to draw definitive conclusions.

Although maternal mobility and peanut ball use during epidural labor appear safe, their effectiveness in improving labor and neonatal outcomes remains inconclusive. Authors consistently call for well-designed randomized controlled trials employing structured and standardized positioning protocols with robust outcome measurement.

At the Women's Wellness and Research Center (WWRC) in Doha, Qatar, epidural analgesia is widely used, particularly among primigravida women. Although peanut birthing balls are available in the Labor and Delivery Unit, their use is not standardized, and maternal positioning is typically guided by individual clinician preference rather than evidence-based protocols. This gap between available resources and optimal practice provides the rationale for the present study.

4. Study Objectives Primary Objective

To evaluate the effect of scheduled maternal position changes using a peanut birthing ball during labor, compared with standard intrapartum care, on maternal and neonatal outcomes among primigravida women receiving epidural analgesia.

Primary maternal outcomes include:

1. Duration of the first and second stages of labor
2. Mode of delivery (spontaneous vaginal, instrumental, or cesarean)
3. Use of intrapartum oxytocin augmentation
4. Estimated blood loss and postpartum hemorrhage
5. Degree of perineal trauma
6. Total hospitalization cost

Primary neonatal outcomes include:

1. Apgar scores at 5 and 10 minutes
2. Admission to the Neonatal Intensive Care Unit (NICU)
3. Birth-related injuries
4. Umbilical cord blood pH

   Secondary Objective

   To examine the association between selected socio-demographic and clinical variables (age, educational level, nationality, employment status, gestational age, and body mass index) and the effect of scheduled maternal positioning using a peanut birthing ball.
5. Study Design and Classification

This study is a prospective, non-invasive, two-arm, parallel-group randomized controlled trial conducted at a single tertiary maternity center.

Participants will be randomized to:

1. Intervention Group: Scheduled maternal position changes using a peanut birthing ball plus standard intrapartum care
2. Control Group: Standard intrapartum care without peanut ball use and without structured positioning

Randomization allows causal assessment of the intervention effect while minimizing bias through standardized protocols.

6. Study Setting and Population

The study will be conducted in the Labor and Delivery Unit of the Women's Wellness and Research Center, Hamad Medical Corporation, Doha, Qatar. The unit manages over 1,300 births per month and follows evidence-based obstetric and midwifery practices.

7. Sample Size and Randomization

Based on prior studies reporting an effect size of approximately 0.66, a sample size of 45 participants per group provides 80% power at a 5% significance level. Allowing for a 20% attrition rate, a total of 110 participants (55 per group) will be recruited.

Randomization will be performed using computer-generated random numbers with allocation concealment. Due to the nature of the intervention, participant and provider blinding is not feasible; however, outcome assessors and data analysts will remain blinded to group allocation.

8. Intervention and Control Conditions Intervention Group

Participants will receive standard intrapartum care plus a structured positioning protocol using a peanut birthing ball following epidural analgesia. Scheduled position changes will include left lateral, right lateral, semi-sitting, and Taylor positions, implemented every 30-60 minutes as clinically appropriate. All positioning will be supervised by trained nursing and midwifery staff.

Control Group

Participants will receive routine intrapartum care following epidural analgesia without the use of a peanut birthing ball or structured positioning schedule.

9. Data Collection and Outcomes

Data will be collected prospectively through real-time observation and electronic medical records. No biological specimens will be collected.

Maternal and neonatal outcomes will be recorded using standardized study forms and entered into a secure electronic database.

10. Data Management and Confidentiality

All participants will be assigned unique study codes. Identifiable information will be stored separately from research data. Electronic data will be password-protected, and paper records will be stored in locked cabinets. Only authorized research personnel will have access to the data.

11. Safety Monitoring

The intervention is considered minimal risk. Continuous maternal and fetal monitoring will be maintained. Any adverse events will be documented and reported according to institutional guidelines.

12. Statistical Analysis

Descriptive statistics will summarize baseline characteristics. Comparative analyses will use appropriate parametric or non-parametric tests. Multivariable models will adjust for potential confounders. Statistical significance will be set at p < 0.05.

13. Ethical Considerations

The study will adhere to the Declaration of Helsinki, Good Clinical Practice guidelines, and institutional regulations. Ethical approval will be obtained prior to study initiation. Participation will be voluntary, and participants may withdraw at any time without impact on clinical care.

14. Funding and Dissemination

Funding is requested from the Hamad Medical Corporation Medical Research Center. Findings will be disseminated through institutional reports, conference presentations, and peer-reviewed publications.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

To be eligible for participation, women must meet all the following criteria:

* Primiparous (first pregnancy resulting in a live birth or stillbirth after 20 weeks of gestation).
* Singleton at gestation.
* Gestational age of the term (37 weeks 0 days to 41 weeks 6 days).
* Admitted to the Labor and Delivery Unit at WWRC in active labor.
* Received epidural analgesia for labor pain management.
* Expected to have a vaginal delivery (e.g., no contraindications for vaginal birth identified at the time of recruitment).
* Able to understand and communicate in Arabic or English.
* Provide written informed consent.

Exclusion Criteria:The birthing ball should NOT be used in any of the following conditions:

1. Obstetric Contraindications (Maternal)

   * Any situation where vaginal birth is not appropriate (e.g., absolute indication for cesarean section)
   * Non-progress of labor requiring immediate intervention
   * Severe pre-eclampsia/eclampsia
   * Active vaginal bleeding of unknown cause
   * Placenta previa (major) or vasa previa
   * Placental abruption (suspected or confirmed)
   * Preterm labor with medical contraindication to ambulation or mobility
   * Ruptured membranes with unstable fetal head (high station) → Risk of cord prolapse
   * Severe maternal exhaustion requiring bed rest
   * Maternal hemodynamic instability
2. Fetal Contraindications

   * Non-reassuring fetal heart rate requiring continuous monitoring (Category II-III tracings)
   * Malpresentation requiring immediate obstetric intervention (e.g., transverse lie)
   * Suspected macrosomia with mechanical obstruction concerns (e.g., cephalopelvic disproportion)
   * Multiple gestation with instability or complications
3. Orthopedic / Musculoskeletal Contraindications

   * Any condition that prevents safe sitting, balancing, or weight-bearing, such as: Severe hips, leg, knee, or pelvic injuries
   * Significant arthritis of the lower limbs or pelvis
   * Recent joint surgery (hip/knee replacement, pelvic repair)
   * Neuromuscular disorders affecting balance (e.g., severe neuropathy)
   * Severe sciatica limiting mobility
   * Poor trunk control or inability to maintain safe seated posture
4. High-Risk Pregnancy Conditions

   * Use of birthing balls is contraindicated if pregnancy is classified as high-risk, including Uncontrolled gestational diabetes and Uncontrolled hypertension
   * Intrauterine growth restriction with required continuous monitoring
   * Polyhydramnios or severe oligohydramnios (risk of cord compression/instability)
   * Preterm premature rupture of membranes (PPROM)
   * History of preterm birth with current instability
   * Any condition requiring bed rest or reduced mobility
5. Safety / Environmental Contraindications

   * Patients are unable to follow instructions or unsteady balance
   * No trained staff available to supervise during labor use Unstable or improperly sized birthing ball

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Females are eligible, as the study involves pregnant, laboring women receiving intrapartum care and first-time full-term pregnancy .
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of First Stage of Labor | 12hours to 16 hours
  Time in minutes from onset of active labor (defined as regular uterine contractions with cervical dilation ≥4-6 cm) to full cervical dilation (10 cm).
Duration of Second Stage of Labor | 2 Hours to 3 Hours
  Time in minutes from full cervical dilation (10 cm) to delivery of the neonate.
Mode of Delivery | At delivery
  Categorized as spontaneous vaginal delivery, instrumental vaginal delivery (forceps or vacuum), or cesarean section.
Use of Oxytocin Augmentation | During labor
  Administration of oxytocin during labor for augmentation of uterine contractions, recorded as yes or no.
Postpartum Hemorrhage | 3 hours after delivery
  Occurrence of postpartum hemorrhage defined as estimated blood loss ≥500 mL following vaginal delivery or ≥1000 mL following cesarean delivery within 24 hours postpartum.
Degree of Perineal Trauma | at time of delivery
  Perineal injury classified as first-degree, second-degree, third-degree (3A, 3B, or 3C), or fourth-degree tear at the time of delivery.
Hospitalization Cost | From admission to discharge
  Total maternal hospitalization cost calculated from admission to discharge based on institutional billing records.
APGAR Score | The Apgar Score is a standardized newborn assessment scale ranging from 0 to 10, with higher scores indicating better neonatal status, assessed at 5 and 10 minutes after delivery.
  Newborn assessment
NICU Admission | 2 hours after delivery
  Number of newborn admissions in NICU
Newborn Birth Injuries | 2 hours from delivery
  Any type of injuries during delivery time

SECONDARY OUTCOMES:
Education Status | 6 months
  Education background of laboring women
BMI | 6 Months
  Body Mass Index
Age | 6 months
  Primiparous Age

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Nather, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Women's Wellness and research center, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared due to the sensitive nature of obstetric and neonatal clinical information and the need to protect participant confidentiality. The dataset contains identifiable intrapartum details that cannot be fully anonymized without compromising data integrity. Additionally, institutional policies at Hamad Medical Corporation restrict the external sharing of raw patient-level data to ensure privacy, data security, and compliance with local regulations. Only aggregated, de-identified results will be shared through publications and presentations.

REFERENCES:
- [Background] 36. Williams, H., Thompson, J., & Lee, A. (2018). The impact of semi-sitting position on labor progression and maternal comfort. Journal of Obstetrics and Gynecology Research, 44(6), 1123-1130.
- [Background] Suraci N, Carr C, Peck J, Hoyos J, Rosen G. Improving labour progression among women with epidural anesthesia following use of a birthing ball: a review of recent literature. J Obstet Gynaecol. 2020 May;40(4):491-494. doi: 10.1080/01443615.2019.1633519. Epub 2019 Sep 3. PMID 31476927
- [Background] Stulz V, Campbell D, Yin B, Al Omari W, Burr R, Reilly H, Lawson K. Using a peanut ball during labour versus not using a peanut ball during labour for women using an epidural: study protocol for a randomised controlled pilot study. Pilot Feasibility Stud. 2018 Oct 4;4:156. doi: 10.1186/s40814-018-0346-9. eCollection 2018. PMID 30305919
- [Background] 29. SÖNMEZ, T., & Apay, S. E. (2023). Effect of Different Birth Balls Used at the First Stage of Labor on Birth Outcomes and Maternal Satisfaction: A Randomized Controlled Trial. Clinical and Experimental Health Sciences, 13(3), 600-607.
- [Background] Salameh KM, Anvar Paraparambil V, Sarfrazul A, Lina Hussain H, Sajid Thyvilayil S, Samer Mahmoud A. Effects of Labor Epidural Analgesia on Short Term Neonatal Morbidity. Int J Womens Health. 2020 Feb 4;12:59-70. doi: 10.2147/IJWH.S228738. eCollection 2020. PMID 32099485
- [Background] 25. Prasad, I. R., & Awasthi, P. (2023). Effectiveness of Squatting Position on the Duration of Labor and Maternal Satisfaction among primigravida Mothers: A Mixed Method Approach. International Journal of Nursing Research, 57-62.
- [Background] Kamath P, Pai M, Shenoy R, Karkada S, D'souza S, Noronha J. Effectiveness of a peanut ball device during labour on maternal and neonatal outcomes: protocol for a randomised controlled trial. F1000Res. 2022 Jun 29;11:717. doi: 10.12688/f1000research.109537.2. eCollection 2022. PMID 36531256
- [Background] Alan Dikmen H, Gonenc IM, Atas AN. Effects of peanut ball use on perceived labor pain, fatigue, and mother's perception of childbirth: a randomized controlled trial. Arch Gynecol Obstet. 2025 Jun;311(6):1579-1589. doi: 10.1007/s00404-024-07656-2. Epub 2024 Aug 5. PMID 39103620
- [Background] 14. Delgado, A. M., da Silva, R. D. C. B., Medeiros, P. J. A., de Souza Melo, R., & de Oliveira, A. L. B. (2022). Peanut ball used for reducing maternal fatigue during labor: protocol for a randomized clinical trial. Research, Society and Development, 11(11),
- [Background] de Verastegui-Martin M, de Paz-Fresneda A, Jimenez-Barbero JA, Jimenez-Ruiz I, Ballesteros Meseguer C. Influence of Laboring People's Mobility and Positional Changes on Birth Outcomes in Low-Dose Epidural Analgesia Labor: A Systematic Review with Meta-Analysis. J Midwifery Womens Health. 2023 Jan;68(1):84-98. doi: 10.1111/jmwh.13446. Epub 2022 Dec 12. PMID 36504479
- [Background] Delgado A, Katz L, Melo RS, Amorim M, Lemos A. Effectiveness of the peanut ball use for women with epidural analgesia in labour: a systematic review and meta-analysis. J Obstet Gynaecol. 2022 Jul;42(5):726-733. doi: 10.1080/01443615.2021.1997959. Epub 2022 Jan 7. PMID 34996318
- [Background] Macena de Almeida ME, Mendes SS, Maria de Vasconcelos Oliveira N, Vasconcelos Neto JA, Lopes LG, Moreira Vasconcelos CT. Peanut Ball Utilization Protocols in Women During Labour and Delivery: An Integrative Review. J Obstet Gynaecol Can. 2023 Nov;45(11):102185. doi: 10.1016/j.jogc.2023.07.005. Epub 2023 Jul 19. PMID 37473916
- [Background] Callahan EC, Lee W, Aleshi P, George RB. Modern labor epidural analgesia: implications for labor outcomes and maternal-fetal health. Am J Obstet Gynecol. 2023 May;228(5S):S1260-S1269. doi: 10.1016/j.ajog.2022.06.017. Epub 2023 Mar 20. PMID 37164496
- [Background] 6. Brown, T., Miller, S., & Davis, K. (2017). Effects of alternating lateral positions on maternal circulation and fetal well-being during labor. Journal of Maternal-Fetal Medicine, 22(4), 210-217
- [Background] 5. Box, M. M. (2023). Implementation and Evaluation of a Peanut Ball Protocol in Laboring Mothers After Epidural Placement (Doctoral dissertation, Southeastern Louisiana University).
- [Background] 3. Ahmed, A. H., Mohmed, A. A., & Fathalla, N. F. (2022). Effect of Peanut Birth Ball on The Progress of Labor and Birth Outcome among Primigravidae. Alexandria Scientific Nursing Journal, 24(4), 91-101.
- [Background] 2. Ahmadpour, A., Bakhshi, S., & Haghani, H. (2020). Use of the peanut ball during labour: A systematic review and meta-analysis. Journal of Clinical Nursing, 29(19-20), 3679-3691. https://doi.org/10.1111/jocn.15338
- [Background] 1. Abdelhady, I. S., Salama, E. I., Ahmed, S. N., Masry, A., & Gad, A. (2023). The Effect of Epidural Analgesia on Maternal and Early Neonatal Outcomes: A Retrospective Cohort Study in Qatar. Journal of Pediatrics, Perinatology and Child Health, 7(1), 55-61.